CLINICAL TRIAL: NCT05360940
Title: Concomitant Infection of Intestinal Parasites and Helicobacter Pylori in Sohag University Hospital
Brief Title: Concomitant Infection of Intestinal Parasites and Helicobacter Pylori
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Nabil Abouzeid, Demonstrator at medical parasitology department at faculty of medicine Sohag university, Sohag University
Other Study IDs: Soh-Med-22-04-15
Record Dates: First submitted 2022-05-01; First posted 2022-05-04 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Dyspepsia Abdominal Burning Pain Diarrhea Dysentery
Keywords: Helicobacter pylori Intestinal Parasites

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: 100 positive stool samples for H.pylori
  Interventions: Diagnostic Test: H.pylori stool antigen rapid test and stool parasitological examination
- B: 100 negative stool samples for H.pylori
  Interventions: Diagnostic Test: H.pylori stool antigen rapid test and stool parasitological examination

INTERVENTIONS:
Diagnostic Test: H.pylori stool antigen rapid test and stool parasitological examination — 200 stool samples ( 100 positive and 100 negative for H.pylori) after performance of H.pylori stool rapid antigen test then parasitological stool examination will be done

SUMMARY:
Intestinal parasitic infections such as Giardia lamblia, Entamoeba histolyica and Enterobius Vermicularis are among the most common infections worldwide.So parasitic infections are considered one of the major health problems in the world especially in developing countries.

Helicobacter pylori is a gram-negative,helical-shaped,motile bacillus bacterium,which colonizes the gastric mucosa.

H.pylori bacterium secretes urease,a special enzyme that converts urea to ammonia.

Ammonia reduces the stomach's acidity .This risk factor allows pathogenic intestinal protozoa such as G.lamblia to take the opportunity to cross through the stomach's increased pH and cause disease.

ELIGIBILITY:
Inclusion Criteria:

* patients complaining of dyspepsia , abdominal burning pain,diarrhea,dysentery,of persons of any age or sex group.

Exclusion Criteria:

* patients taking antibiotics within the previous four weeks, proton pump inhibitors within the previous two weeks, or anti-parasitic drugs within the previous two weeks.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Samples will be collected from outpatients complaining of dyspepsia, abdominal burning pain, diarrhea,and dysentery with persons of any age or sex groups from different locations (cities and villages)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Compare the prevalence of intestinal parasitic infections among positive and negative H.pylori infected outpatients in Sohag University Hospital | 18 weeks following the start point of the study
  Collection of 200 stool samples (100 positive and 100 negative for H.pylori) then parasitological examination done for all samples

SECONDARY OUTCOMES:
Evaluate the prevalence of intestinal parasitic infection among H.pylori infected outpatients in Sohag University Hospital | 18 weeks following the start point of the study
  Macroscopic and microscopic examination of 100 positive H.pylori stool samples

CONTACTS AND LOCATIONS:
Locations (1):
- Asmaa Nabil Abouzeid, Sohag, Egypt